CLINICAL TRIAL: NCT07387367
Title: A Phase 3, Multicenter, Prospective, Randomized, Open-label Efficacy and Safety Study of Intravenous Brincidofovir Versus Intravenous Cidofovir for Treatment of Adenovirus Infection in Pediatric and Adult Subjects After Allogeneic Hematopoietic Cell Transplantation (Allo-HCT)
Brief Title: A Phase 3 Trial to Compare IV BCV Versus IV CDV for Treatment of Adenovirus Infection After Allo-HCT
Acronym: ENOVIA
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: SymBio Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BCV-PA02
Record Dates: First submitted 2026-01-20; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Adenovirus Infections
Keywords: Brincidofovir; Cidofovir; Adenovirus; allo-HCT; BCV-PA02; ENOVIA
MeSH Terms: conditions — Adenoviridae Infections | interventions — Cidofovir; brincidofovir

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IV BCV (Experimental)
  Interventions: Drug: Brincidofovir
- IV CDV (Active Comparator)
  Interventions: Drug: cidofovir

INTERVENTIONS:
Drug: cidofovir — CDV does not have a labeled indication for treating Adenovirus infection. CDV will be administered according to local guidelines and institutional standard of care practice.
  Other Names: IV CDV
  Arms: IV CDV
Drug: Brincidofovir — Intravenous
  Other Names: SyB V-1901
  Arms: IV BCV

SUMMARY:
This randomized, open-label, parallel group, two-arm, multi-center assessment will compare IV BCV with IV CDV in adult and pediatric allogeneic HCT recipients with AdV viremia. A virologic response-driven approach to duration of treatment will be evaluated, in which randomized subjects are treated with either BCV or CDV until AdV viremia is confirmed as undetectable or until a maximum of 12 weeks of therapy, whichever occurs first. All subjects will be followed for a total of 24 weeks post-randomization, regardless of treatment assignment. Subjects will be assessed on a weekly basis through the end of treatment visit (EOT). Additional assessments will be performed at the test of cure (TOC) visit, which is 4 weeks after the last dose of study drug and at Weeks 12 and 24 post W1D1.

DETAILED DESCRIPTION:
This Phase 3 multi-center, randomized, open-label study will assess efficacy of IV BCV, compared to IV CDV, in allo-HCT subjects with AdV viremia. Randomized subjects will be treated for up to a maximum of 12 weeks of therapy for both arms. Primary efficacy assessment will be performed at W5D1. Consistent with ECIL guidelines for high-risk patients, AdV viremia will be assessed weekly. Subjects randomized to receive BCV or CDV are treated until AdV DNA is confirmed to be undetectable in plasma for two consecutive tests 7 days apart, or until Week 12 post W1D1, whichever occurs first. Subjects will continue BCV or CDV as long as AdV viremia is detectable, contingent on tolerability, until viremia clears, or the subject reaches a maximum duration of 12 weeks of study drug treatment.

Subjects will receive assigned randomized therapy until time of AdV virological success plus 2 weeks, for up to a maximum of 12 weeks. All subjects will be followed through 24 weeks. All study visits and follow-up assessments must be completed regardless of the study drug treatment duration. All subjects are considered on study through the Week 24 follow-up visit.

For subjects who achieve virological success from their initial randomized study drug treatment and experience an AdV viremia recurrence, repeat treatment with their randomized study drug is allowed. There is no cross-over study drug treatment allowed in this study and subjects can only receive retreatment with their randomized study drug.

Subjects who stop study drug therapy due to confirmed undetectable AdV viremia may re-initiate study drug treatment if AdV viremia is subsequently confirmed at ≥ 1000 IU/mL by the designated central virology laboratory (recurrence). For the purposes of re-initiating study drug therapy, "confirmed viremia ≥ 1000 IU/mL" is defined as two consecutive results ≥ 1000 IU/mL from the designated central laboratory, with the second sample drawn at least 48 hours after the first sample.

Subjects who permanently discontinue study drug therapy for toxicity reasons are not eligible to re-initiate study drug dosing. Study procedures are to be followed during these Retreatment visits as applicable for BCV and CDV outlined in the schedule of assessments (SOA).

An independent Data Safety Monitoring Board (DSMB) will review accumulated safety data for this study when total combined enrollment in both arms is approximately 25% (45 subjects) and 50% (90 subjects). They will also review adverse events on an ongoing basis. They will make recommendations to the Sponsor based on review of these safety data. Further details regarding data safety monitoring guidelines will be included in the DSMB Charter. The DSMB will make determinations regarding continued enrolment and/or stopping the study for safety reasons.

An Endpoint Adjudication Committee (EAC) will be convened to evaluate baseline diagnosis and AdV disease clinical response as outlined in the EAC charter.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female, post-allo HCT within last 180 days, aged 2 months and older at time of signing informed consent form.
2. Subject/Guardian willing and able to understand and provide written informed consent to participate in the study.
3. In the investigator's judgement, the subject's clinical condition justifies treatment with IV BCV or IV CDV for AdV infection.
4. Has adenoviremia, based on any of:

   * AdV viremia DNA ≥10,000 IU/mL, OR
   * Two consecutive and rising AdV viremia DNA results of ≥1,000 IU/mL at screening, OR
   * AdV viremia DNA of ≥1,000 IU/mL, AND

1. Lymphocyte count <180/mm3, OR 2. Received T cell depletion, cord blood, or haploidentical transplant, OR 3. prior alemtuzumab, OR 4. anti-thymocyte globulin (ATG)

Exclusion Criteria:

1. Subject received an allo-HCT with a matched sibling donor
2. Subject received more than 5 mg/kg of CDV for any reason in the 21 days prior to first dose of study drug.
3. Subject is allergic or hypersensitive to IV BCV or IV CDV or any of their components.
4. Subject received anti-AdV-specific cell-based therapy within 3 weeks prior to W1D1 or an anti-AdV vaccine at any time.
5. Subject has participated in any other investigational study within 30 days (or within 5.5 half-lives of the investigational product, whichever is longer) before signing the informed consent form (ICF), is currently participating in another interventional treatment trial with an investigational agent or is using an investigational device at the time of Screening.

Min Age: 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
To assess efficacy of intravenous (IV) brincidofovir (BCV), compared with IV cidofovir (CDV), in subjects after allo-HCT with adenovirus (AdV) viremia. | Week (W) 5 Day (D) 1.
  The primary efficacy endpoint is defined as AdV virological success at W5D1.
  -Proportion of subjects with AdV virological success

SECONDARY OUTCOMES:
To assess the efficacy and safety of IV BCV, and IV CDV, in subjects after allo-HCT with AdV viremia. | Test Of Cure (Last Dose + 30 days)
  The proportion of subjects with overall success, as adjuducated by the EAC
To assess the efficacy and safety of IV BCV, and IV CDV, in subjects after allo-HCT with AdV viremia. | Week 1 Day 1 Through End Of Study (Week 24).
  Incidence and severity of treatment-emergent adverse events (TEAEs).
To assess the efficacy and safety of IV BCV, and IV CDV, in subjects after allo-HCT with AdV viremia. | Week 5 Day 1, Last Dose + 4 Days, Last Dose + 30 days, Week 12, and Week 24.
  All cause mortality
BCV Plasma Concentrations will be collected, measured and reported | Plasma samples will be collected at Week 1 Day 1, and Week 5 Day 1
  The drug level (BCV) in plasma will be measured and used to examine the variability in drug concentrations among patients within the study population (i.e., population pharmacokinetics analysis).

CONTACTS AND LOCATIONS:
Overall Officials: Nkechi Azie, Study Director — SymBio Pharmaceuticals
Locations (61):
- United States (26):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - City of Hope, Duarte, California
  - University of California Davis, Sacramento, California
  - Rady Children's Hospital, San Diego, California
  - Children's Hospital Colorado-Center for Cancer and Blood Disorders, Aurora, Colorado
  - Children's National Hospital, Washington D.C., District of Columbia
  - Children's Healthcare of Atlanta/Emory, Atlanta, Georgia
  - Ann and Robert H Lure Children's Hospital, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Dana-Farber Cancer Institute-Brighman and Women's, Boston, Massachusetts
  - Dana-Farber/Boston Children's Cancer and Blood Disorders Center, Boston, Massachusetts
  - Helen Devos Children's Hospital / Michigan State University, Grand Rapids, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - St Louis Children's Hospital - Barnes Jewish Hospital, St Louis, Missouri
  - University of Nebraska, Omaha, Nebraska
  - Joseph M Sanzari Children's Hospital, Hackensack, New Jersey
  - Cohen Children's Medical Center, New Hyde Park, New York
  - Weill Cornell Medicine, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pittsburg Medical Center Children's Hospital, Pittsburgh, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Seattle Children's Hospital, Seattle, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
- St. Anna Kinderspital- Childrens Hospital, Vienna, Austria
- Leuven, University Hospital Gasthuisberg, Leuven, Belgium
- Canada (3):
  - Alberta Children's Hospital University of Calgary, Calgary
  - CHU Sainte Justine Hospital, Montreal
  - The Hospital for Sick Children, Toronto
- France (3):
  - Hôpital Saint-Louis, Paris
  - Necker Hospital, Paris
  - Robert-Debré Hospital, APHP Nord Université de Paris Cité., Paris
- Germany (7):
  - Charité University Hospital, Berlin
  - Essen University Hospital, Essen
  - University Hospital Frankfurt, am Main, Frankfurt
  - University Medical Center Hamburg-Eppendorf (UKE), Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - University Children's Hospital, Münster
  - Kinderheilkunde I | Universitätsklinikum Tübingen, Tübingen
- Italy (5):
  - Istituto Giannina Gaslini, Genova
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Perugia Hospital, Perugia
  - Ospedale Pediatrico Bambino Gesu', Rome
  - IRCCS San Raffaele Hospital, San Raffaele
- Netherlands (2):
  - Leiden Unviversity Medical Center, Leiden
  - Princess Maxima Center & UMC Utrecht, Utrecht
- Instituto Português de Oncologia do Porto (IPO Porto) Francisco Gentil, EPE, Porto, Portugal
- Spain (3):
  - Vall d'Hebron University Hospital, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Clinica Universidad de Navarra, Pamplona
- Karolinska University Hospital, Stockholm, Sweden
- United Kingdom (8):
  - Birmingham Women's and Children's Hospital, Birmingham
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - Great Ormond Street Hospital for Children, London
  - University College London Hospitals NHS Foundation Trust, London
  - Royal Manchester Children's Hospital, Manchester
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust - Freeman Hospital, Newcastle upon Tyne
  - Sheffield Children's Hospital, Sheffield
  - Royal Marsden Hospital, Sutton

IPD SHARING:
Plan to Share IPD: No